CLINICAL TRIAL: NCT03184597
Title: HLA Screening in Reducing the Risk of Antiepileptic Drug-induced Cutaneous Adverse Reactions: a Multicenter Clinical Study
Brief Title: HLA Screening in Reducing the Risk of Antiepileptic Drug-induced Cutaneous Adverse Reactions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Guangzhou First People's Hospital (Other); West China Hospital (Other); Guangdong Provincial People's Hospital (Other); First Affiliated Hospital of Jinan University (Other); Guangdong 999 Brain Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Wuhan Women and Children's Medical Center (Other); First People's Hospital, Shunde China (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-hs-30
Record Dates: First submitted 2017-06-09; First posted 2017-06-12 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Epilepsy; Neuropathy; Psychiatric Illness; Blepharospasm
Keywords: HLA screening; SJS/TEN; MPE; AEDs
MeSH Terms: conditions — Epilepsy; Mental Disorders; Blepharospasm; Stevens-Johnson Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group with two strong risk factors (Experimental): When HLA screening before commencing aromatic AEDs shows positive for both HLA-A*24:02 and HLA-B*15:02 in a patient, aromatic AEDs were not administrated for this patient.
  Interventions: Diagnostic Test: HLA screening before commencing aromatic AEDs
- Group with one strong risk factors (Experimental): When HLA screening before commencing aromatic AEDs shows positive for HLA-B*15:02, carbamazepine (CBZ) was not administrated, and other aromatic AEDs were prescribed with caution or avoided if alternative non-aromatic AEDs can be prescribed instead.
  When HLA screening before commencing aromatic AEDs shows positive for HLA-B*15:01 or HLA-A*24:02, aromatic AEDs were prescribed with caution or avoided if alternative non-aromatic AEDs can be prescribed instead.
  Interventions: Diagnostic Test: HLA screening before commencing aromatic AEDs
- Group with one potential risk factors (Experimental): When HLA screening before commencing aromatic AEDs shows positive for any potential risk allele such as HLA-B*15:11, HLA-A*02:01and HLA-DRB1*01:01, aromatic AEDs were prescribed with caution or avoided if alternative non-aromatic AEDs can be prescribed instead.
  Interventions: Diagnostic Test: HLA screening before commencing aromatic AEDs
- Group without known risk factors (Experimental): When HLA screening before commencing aromatic AEDs shows negative for any known HLA risk allele , aromatic AEDs was administrated to these patients.
  Interventions: Diagnostic Test: HLA screening before commencing aromatic AEDs

INTERVENTIONS:
Diagnostic Test: HLA screening before commencing aromatic AEDs — When the risk HLA alleles are tested positive for the patients, aromatic AEDs were avoided or administrated with caution according to the risk level.

SUMMARY:
Cutaneous adverse drug reactions (cADRs) include mild maculopapular exanthema (MPE) and severe cutaneous reactions such as hypersensitivity syndrome, Stevens-Johnson syndrome (SJS), and toxic epidermal necrolysis (TEN). cADRs are considered as a major public health issue because of their potentially life-threatening morbidity, especially severe cutaneous reactions. The incidence of SJS/TEN is estimated to vary from 1 in 1,000 to 10,000 drug exposures, and its mortality is as high as 35%. Antiepileptic drugs (AEDs), particularly those with aromatic ring structures such as carbamazepine (CBZ), oxcarbazepine (OXC), lamotrigine (LTG), phenobarbital (PB), and phenytoin (PHT), are among the most common causes of severe cutaneous reactions. The incidence of AED-induced SJS was estimated as 0.2% and all cases occurred in individuals receiving aromatic AEDs.

Previous studies have validated that the human leukocyte antigen (HLA) allele HLA-B*15:02 is strongly associated with CBZ-induced SJS/TEN in southern Han Chinese and populations in southeast Asia. Our recent studies indicated that HLA-A*24:02 is a common genetic risk factor for CBZ-, LTG-, and PHT-induced SJS/TEN. It is also associated with MPE. Additionally, another four alleles, including HLA-B*15:01, HLA-B*15:11, HLA-A*02:01,and HLA-DRB1*01:01, were showed to be potential risk factors for aromatic AEDs-induced SJS/TEN. In 2007, the US Food and Drug Administration issued the safety alert that recommended HLA-B*15:02 screening for people with Asian ancestry before starting CBZ, and avoidance of the drug if the test is positive. Subsequent studies from Taiwan, Hong Kong and Thailand demonstrated that HLA-B*15:02 screening before commencing CBZ can significantly reduce the incidence of CBZ-induced SJS/TEN. However, the overall incidence of AEDs-induced SJS/TEN remained unchanged in Hong Kong, as PHT-induced SJS/TEN increased when CBZ-SJS/TEN decreased. Moreover, no study focuses on the incidences of AEDs-induced cADRs with and without HLA screening before commencing aromatic AEDs. Therefore, we are planning to conduct a multicenter prospective study to examine the reduction of AEDs-induced cADRs after the HLA screening prior to the beginning of aromatic AEDs administration.

DETAILED DESCRIPTION:
In this prospective study, 4000 or more patients from multicenters in southern China will be recruited. A HLA screening will be conducted before these patients start aromatic AEDs treatments. According to the HLA genotype, these patients will be divided into four groups that are three positive groups with different risk alleles and one negative group with no known risk allele. Aromatic AEDs were avoided or administrated with caution according to the risk level in the three positive groups, while they can be prescribed in the negative group. The effectiveness of HLA screening prior to the beginning of aromatic AEDs administration will be observed by the reduction of overall incidence of AEDs-induced cADRs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are going to receive a kind of aromatic AEDs including CBZ, OXC, LTG, PHT, and PB as a new therapy. An AED was deemed newly commenced if there was no record of its prescription in at least the previous 12 months.
2. Ethnic Han Chinese. None of the biological grandparents of the participants were from other races.

Exclusion Criteria:

1. individuals who are not of Han Chinese descent.
2. individuals who had undergone bone marrow transplantation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
AEDs-induced cADRs incidence | 3 months
  the incidence of AEDs-induced cADRs within the first 3 months of commencing an aromatic AED

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Ping Liao, M.D.,Ph.D., Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical Universty, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The clinical data and HLA genotype of the participant will be shared in the collaborators
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 2017 July - 2021 July

REFERENCES:
- [Background] Shi YW, Min FL, Zhou D, Qin B, Wang J, Hu FY, Cheung YK, Zhou JH, Hu XS, Zhou JQ, Zhou LM, Zheng ZZ, Pan J, He N, Liu ZS, Hou YQ, Lim KS, Ou YM, Hui-Ping Khor A, Ng CC, Mao BJ, Liu XR, Li BM, Kuan YY, Yi YH, He XL, Deng XY, Su T, Kwan P, Liao WP. HLA-A*24:02 as a common risk factor for antiepileptic drug-induced cutaneous adverse reactions. Neurology. 2017 Jun 6;88(23):2183-2191. doi: 10.1212/WNL.0000000000004008. Epub 2017 May 5. PMID 28476759
- [Background] Shi YW, Min FL, Qin B, Zou X, Liu XR, Gao MM, Wang Q, Zhou JQ, Liao WP. Association between HLA and Stevens-Johnson syndrome induced by carbamazepine in Southern Han Chinese: genetic markers besides B*1502? Basic Clin Pharmacol Toxicol. 2012 Jul;111(1):58-64. doi: 10.1111/j.1742-7843.2012.00868.x. Epub 2012 Mar 17. PMID 22348435
- [Background] Shi YW, Min FL, Liu XR, Zan LX, Gao MM, Yu MJ, Liao WP. Hla-B alleles and lamotrigine-induced cutaneous adverse drug reactions in the Han Chinese population. Basic Clin Pharmacol Toxicol. 2011 Jul;109(1):42-6. doi: 10.1111/j.1742-7843.2011.00681.x. Epub 2011 Mar 16. PMID 21306565
- [Background] Chen P, Lin JJ, Lu CS, Ong CT, Hsieh PF, Yang CC, Tai CT, Wu SL, Lu CH, Hsu YC, Yu HY, Ro LS, Lu CT, Chu CC, Tsai JJ, Su YH, Lan SH, Sung SF, Lin SY, Chuang HP, Huang LC, Chen YJ, Tsai PJ, Liao HT, Lin YH, Chen CH, Chung WH, Hung SI, Wu JY, Chang CF, Chen L, Chen YT, Shen CY; Taiwan SJS Consortium. Carbamazepine-induced toxic effects and HLA-B*1502 screening in Taiwan. N Engl J Med. 2011 Mar 24;364(12):1126-33. doi: 10.1056/NEJMoa1009717. PMID 21428768
- [Background] Chen Z, Liew D, Kwan P. Effects of a HLA-B*15:02 screening policy on antiepileptic drug use and severe skin reactions. Neurology. 2014 Nov 25;83(22):2077-84. doi: 10.1212/WNL.0000000000001034. Epub 2014 Oct 29. PMID 25355835
- [Background] Rattanavipapong W, Koopitakkajorn T, Praditsitthikorn N, Mahasirimongkol S, Teerawattananon Y. Economic evaluation of HLA-B*15:02 screening for carbamazepine-induced severe adverse drug reactions in Thailand. Epilepsia. 2013 Sep;54(9):1628-38. doi: 10.1111/epi.12325. Epub 2013 Jul 29. PMID 23895569
- [Background] Chen Z, Liew D, Kwan P. Real-world cost-effectiveness of pharmacogenetic screening for epilepsy treatment. Neurology. 2016 Mar 22;86(12):1086-94. doi: 10.1212/WNL.0000000000002484. Epub 2016 Feb 17. PMID 26888992